CLINICAL TRIAL: NCT04380220
Title: Coagulation/Complement Activation and Cerebral Hypoperfusion in Relapsing-remitting Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Roma La Sapienza (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Tatiana Koudriavtseva, Principal Investigator, Regina Elena Cancer Institute
Other Study IDs: 972/17; PE-2013-02357745 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis; Relapse
Keywords: multiple sclerosis; relapse; coagulation; complement; cerebral blood flow
MeSH Terms: conditions — Multiple Sclerosis; Recurrence; Thrombosis | interventions — Blood Specimen Collection; Partial Thromboplastin Time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Serum/plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Relapsing MS patients: Patients diagnosed with relapsing-remitting multiple sclerosis and in relapse, untreated or treated with only immunomodulatory therapy.
  Interventions: Diagnostic Test: Blood samples and processing
- Remitting MS patients: Patients diagnosed with relapsing-remitting multiple sclerosis and in remission, untreated or treated with only immunomodulatory therapy.
  Interventions: Diagnostic Test: Blood samples and processing
- Healthy controls: Age- and sex-matched healthy control subjects.
  Interventions: Diagnostic Test: Blood samples and processing

INTERVENTIONS:
Diagnostic Test: Blood samples and processing — DSC perfusion technique at 3.0-T MRI only in MS patients
  Other Names: complement C3, C4, C4a, C9, fibrinogen, factor VIII and X, D-dimer, protein C, protein S, antithrombin, aPTT, factor II, v-Willebrand factor, thrombomodulin, Endothelial Protein C Receptor

SUMMARY:
This is a multi-center, prospective, controlled study. MS patients (1° group: 30 patients in relapse; 2° group: 30 patients in remission) and age/sex-matched healthy controls (3° group: 30 subjects) will be enrolled in the study. Patients' disability level will be evaluated by EDSS and MSFC.

Patients and controls will be tested for either coagulation/complement (C3, C4, C4a, C9, fibrinogen, factor VIII and X, D-dimer, protein C, protein S, antithrombin, factor II, aPTT, von-Willebrand factor), soluble markers of endothelial damage (thrombomodulin, Endothelial Protein C Receptor), antiphospholipid antibodies, lupus anticoagulant, complete blood count, viral serological assays or microRNA microarray.

Patients will undergo dynamic susceptibility contrast-enhanced MRI using a 3.0-T scanner to evaluate CBF, CBV, MTT, lesion number and volume.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with relapsing-remitting multiple sclerosis, untreated or treated with only immunomodulatory therapy, in relapse o in remission

Exclusion Criteria:

* pregnant, with any neoplastic, hematologic, thyroid, metabolic, thrombotic or autoimmune disease, drug or alcohol addicted, treated with immunosuppressive drugs, steroids o any medication interfering with coagulation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Relapsing-remitting multiple sclerosis patients and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
plasma concentration of coagulation factor | through study completion, an average of 1 year
  Factor VIII (%)
plasma concentration of coagulation factor | through study completion, an average of 1 year
  Factor X (%)
plasma concentration of coagulation factor | through study completion, an average of 1 year
  D-dimer (ng/ml)
plasma concentration of coagulation factor | through study completion, an average of 1 year
  Protein C (%)
plasma concentration of coagulation factor | through study completion, an average of 1 year
  Protein S (%)
plasma concentration of coagulation factor | through study completion, an average of 1 year
  Fibrinogen (mg/dl)
plasma concentration of coagulation factor | through study completion, an average of 1 year
  complement (mg/dl)

SECONDARY OUTCOMES:
Brain MRI hemodynamic changes at DSC 3.0-T MRI | through study completion, an average of 1 year
  cerebral blood flow
Brain MRI hemodynamic changes at DSC 3.0-T MRI | through study completion, an average of 1 year
  cerebral blood volume
Brain MRI hemodynamic changes at DSC 3.0-T MRI | through study completion, an average of 1 year
  mean transit time

CONTACTS AND LOCATIONS:
Locations (3):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Italy (2):
  - IRCCS Regina Elena National Cancer Institute, Rome
  - University of Rome Sapienza, Rome

REFERENCES:
- [Derived] Koudriavtseva T, Lorenzano S, Cellerino M, Truglio M, Fiorelli M, Lapucci C, D'Agosto G, Conti L, Stefanile A, Zannino S, Filippi MM, Cortese A, Piantadosi C, Maschio M, Maialetti A, Galie E, Salvetti M, Inglese M. Tissue factor as a potential coagulative/vascular marker in relapsing-remitting multiple sclerosis. Front Immunol. 2023 Jul 31;14:1226616. doi: 10.3389/fimmu.2023.1226616. eCollection 2023. PMID 37583699
- [Derived] Koudriavtseva T, Stefanile A, Fiorelli M, Lapucci C, Lorenzano S, Zannino S, Conti L, D'Agosto G, Pimpinelli F, Di Domenico EG, Mandoj C, Giannarelli D, Donzelli S, Blandino G, Salvetti M, Inglese M. Coagulation/Complement Activation and Cerebral Hypoperfusion in Relapsing-Remitting Multiple Sclerosis. Front Immunol. 2020 Oct 27;11:548604. doi: 10.3389/fimmu.2020.548604. eCollection 2020. PMID 33193314